CLINICAL TRIAL: NCT01195324
Title: An Open-Label Drug Interaction Study to Assess the Pharmacokinetics and Pharmacodynamics of Warfarin When Administered Alone and in Combination With Multiple-Dose JNJ-28431754 (Canagliflozin) in Healthy Male and Female Subjects
Brief Title: A Drug Interaction Study of Warfarin and Canagliflozin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR017440
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Canagliflozin (JNJ-28431754); Warfarin; Pharmacokinetic; Pharmacodynamic; Prothrombin time (PT); International normalized ratio (INR)
MeSH Terms: interventions — Canagliflozin; Warfarin

ARMS (2):
- 001 (Experimental): Canagliflozin/Warfarin Treatment A: Tablets oral canagliflozin 300 mg once daily for 12 days and canagliflozin 300 mg + warfarin 30 mg single dose on Day 6 followed 14 days later by Treatment B: Tablets oral warfarin 30 mg single dose on Day 1
  Interventions: Drug: Canagliflozin/Warfarin
- 002 (Experimental): Canagliflozin/Warfarin Treatment B: Tablets oral warfarin 30 mg single dose on Day 1 followed 14 days later by Treatment A: Tablets oral canagliflozin 300 mg once daily for 12 days and canagliflozin 300 mg + warfarin 30 mg single dose on Day 6
  Interventions: Drug: Canagliflozin/Warfarin

INTERVENTIONS:
Drug: Canagliflozin/Warfarin — Treatment A: Tablets, oral, canagliflozin 300 mg, once daily for 12 days and canagliflozin 300 mg + warfarin 30 mg, single dose on Day 6 followed 14 days later by Treatment B: Tablets, oral, warfarin 30 mg, single dose on Day 1
  Arms: 001
Drug: Canagliflozin/Warfarin — Treatment B: Tablets, oral, warfarin 30 mg, single dose on Day 1 followed 14 days later by Treatment A: Tablets, oral, canagliflozin 300 mg, once daily for 12 days and canagliflozin 300 mg + warfarin 30 mg, single dose on Day 6
  Arms: 002

SUMMARY:
The purpose of the study is to assess the effect of multiple oral doses of canagliflozin on a single oral dose of warfarin.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center study of canagliflozin (JNJ-28431754) and warfarin in healthy adult volunteers. Canagliflozin is a drug currently under development to lower blood sugar levels in patients with type 2 diabetes mellitus and warfarin is an approved anticoagulant (ie, a drug that stops blood from clotting). After an overnight fast (without eating food) of at least 10 hours, volunteers will receive Sequence 1 (canagliflozin 300 mg, orally, once daily on Days 1-12 with a single, oral 30 mg dose of warfarin on Day 6 [Treatment A] followed 14 days later by a single, oral 30 mg dose of warfarin on Day 1 [Treatment B]) OR Sequence 2 (Treatment B followed 14 days later by Treatment A).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index between 18 and 30 kg/m

Exclusion Criteria:

* Any blood coagulation disorder determined to be clinically relevant by the Investigator
* Medications known to affect coagulation taken within 7 to 14 days of study entry

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | At protocol-specified times during Treatment A on Days 1 through 12.
Plasma concentrations of warfarin | At protocol specified times during Treatment A on Days 6 through 13
Plasma concentrations of warfarin | At protocol specified times during Treatment B on Days 1 through 8
Measurement of Prothrombin time (PT) to assess the international normalized ratio (INR) | At protocol-specified times during Treatment A on Days 6 through 13
Measurement of PT to assess the INR | At protocol-specified time points during Treatment B on Days 1 through 8

SECONDARY OUTCOMES:
The number and type of adverse events reported | Day 1 of Treatment A through 10 days after Day 8 of Treatment B
The number and type of adverse events reported | Day 1 of Treatment B through 10 days after Day 13 of Treatment A

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Vaccaro N, Bernard A, Skee D, Mamidi RN, Tian H, Weiner S, Stieltjes H, Sha S, Rothenberg P. Effect of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on the pharmacokinetics of oral contraceptives, warfarin, and digoxin in healthy participants. Int J Clin Pharmacol Ther. 2015 Jan;53(1):41-53. doi: 10.5414/CP202157. PMID 25345427